CLINICAL TRIAL: NCT06550908
Title: Training Physicians to Differentiate the Paris Classification Using Artificial Colon Polyp Images
Acronym: LUTETIA2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022120701-2
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Colonic Polyp; Colon Adenoma
Keywords: Colonoscopy
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training with real images (Active Comparator): Physicians train using the Paris classification with real colon polyp images
  Interventions: Other: Lutetia Training Plattform - real images
- Training with artificial images (Experimental): Physicians train using the Paris classification with artificial colon polyp images
  Interventions: Other: Lutetia Training Plattform - artifical images

INTERVENTIONS:
Other: Lutetia Training Plattform - real images — Training platform Lutetia offers training the Paris classification using real images of colon polyps.
  Arms: Training with real images
Other: Lutetia Training Plattform - artifical images — Training platform Lutetia offers training the Paris classification using artificial images of colon polyps.
  Arms: Training with artificial images

SUMMARY:
Training in endoscopy is essential for the early detection of precursors of colorectal cancer. Up to now, this training has been carried out with image collections of findings and in practice when working on patients. The investigators want to use artificial intelligence (AI) to better train doctors to recognise these precursors. By using generative AI, the investigators were able to create realistic images that comply with data protection regulations and whose content can be predefined. Parts of the image can also be regenerated so that it is possible to create different precancerous stages in the same place in the image.

In this study the investigators want to train physicians using real images or artificial images in order to compare which version helps classify polyps better.

ELIGIBILITY:
Inclusion Criteria:

* Physicians with or without experience in colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy for Paris classification | 9 months
  Ability to correctly classify colonic polyps using the Paris classification

SECONDARY OUTCOMES:
Range of misclassifications for Paris classification | 9 months
  Number of misclassification categorizes (eg 1-4)
Influence of endoscopy experience on accuracy for correct Paris classification | 9 months
  Influence of endoscopy experience measured in number of perfomed colonoscopies on accuracy for correct Paris classification
Influence of time to complete course on accuracy for correct Paris classification | 9 months
  Influence of time to complete course measured in days on accuracy for correct Paris classification
Influence regular usage of Paris classification on accuracy for correct Paris classification | 9 months
  Influence regular usage of Paris classification (yes/no) on accuracy for correct Paris classification

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hann, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- University hospital Würzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No